CLINICAL TRIAL: NCT04630379
Title: Pilot Study of Early Integration of Palliative Care Using the BEACON PROQOL in Patients With High Grade Glioma and Their Caregivers
Brief Title: Early Integration of Palliative Care Using the BEACON PROQOL in Patients With High Grade Glioma and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alyx Porter, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-011342; NCI-2020-07998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-011342 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma; Malignant Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (visit with neuro-oncologist) (Experimental): Patients and primary caregiver complete the BEACON PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist monthly for 6 months to address concerns that are identified via the survey and the domain of concern identified by patient and caregiver.
  Interventions: Other: Quality-of-Life Assessment; Other: Supportive Care; Other: Survey Administration
- Group B (visit with neuro-oncologist and palliative care team) (Experimental): Patients and primary caregiver complete the BEACON PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist and palliative care team monthly for 6 months to address concerns that are identified by the survey and domains of concerns. Caregivers also attend support sessions led by a social worker monthly for 6 months.
  Interventions: Other: Palliative Therapy; Other: Quality-of-Life Assessment; Other: Supportive Care; Other: Survey Administration
- Group C (visit with neuro-oncologist, palliative care team) (Active Comparator): Patients and primary caregiver complete quality of life portion of the BEACON PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist monthly for 6 months and address important concerns that come up on the survey. Patients may also receive palliative care consultation as deemed appropriate by the neuro-oncologist.
  Interventions: Other: Palliative Therapy; Other: Quality-of-Life Assessment; Other: Supportive Care; Other: Survey Administration

INTERVENTIONS:
Other: Palliative Therapy — Visit with palliative care team
  Other Names: Comfort Care; PA-Palliative Therapy; palliation; Palliative; Palliative Care; Palliative Treatment; Symptom Management; Symptoms Management
  Arms: Group B (visit with neuro-oncologist and palliative care team); Group C (visit with neuro-oncologist, palliative care team)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Supportive Care — Visit with neuro-oncologist
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
Other: Survey Administration — Complete survey

SUMMARY:
This trial assesses the quality of life in patients with high grade glioma and their caregivers using a questionnaire called the Beacon Patient Related Outcomes Quality of Life (PROQOL). Knowledge gained from this trial may help researchers find out if early integration of palliative care will lead to improvement in quality of life for both patients and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess feasibility of intra-office Beacon Patient Related Outcomes Quality of Life Scale (PROQOL) assessment of patient and caregiver.

II. Assess feasibility of routine (monthly) visits with palliative care specialists.

III. Evaluate if overall quality of life of patients with high grade glioma and their caregivers improves with identifying and addressing symptoms and psychosocial concerns identified through the PROQOL tool.

IV. Evaluate if overall quality of life of patients with high grade glioma improves further with early integration of palliative care.

V. Evaluate if overall quality of life of primary caregivers improves with early integration of palliative care.

VI. Compare patient's perception and understanding of disease severity and prognosis with that of the caregivers, and with that of the clinicians.

VII. Evaluate variance in prognosis between the neurooncologist and palliative care specialist.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP A: Patients and primary caregiver complete the Beacon PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist monthly for 6 months to address concerns that are identified via the survey and the domain of concern identified by patient and caregiver.

GROUP B: Patients and primary caregiver complete the Beacon PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist and palliative care team monthly for 6 months to address concerns that are identified by the survey and domains of concerns. Caregivers also attend support sessions led by a social worker monthly for 6 months.

GROUP C: Patients and primary caregiver complete quality of life portion of the Beacon PROQOL survey before each visit. Patients then receive standard of care for high grade glioma consisting of visits with neuro-oncologist monthly for 6 months and address important concerns that come up on the survey. Patients may also receive palliative care consultation as deemed appropriate by the neuro-oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Adults with pathology confirmed high grade glioma, graded as World Health Organization (WHO) grade III and IV
* Ability to use a tablet
* Able to adhere to completing surveys at study visits
* English speaking
* Has a caregiver that has provided oral consent to participate in this study
* Insurance accepted at Mayo Clinic Arizona

Exclusion Criteria:

* Inability to use a tablet
* Inability to adhere to completing surveys at monthly visits
* Unable to speak English
* Lack of a caregiver
* Insurance not accepted at Mayo Clinic Arizona

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in feasibility of using the Beacon Patient Reported Outcomes Quality of Life Scale (PROQOL) | monthly for six months
  Patients will be randomized to 3 groups - Control (standard of care); Arm A (PROQOL + standard of care); Arm B (early palliative care + Arm A). Feasibility of conducting the assessment at monthly visits for each patient/caregiver cluster, along with early involvement of palliative care, will be assessed.
Change in feasibility of using a single question to assess prognostic understanding in patients, caregivers, and clinicians | monthly for 6 months
  At each visit, patients, their caregivers, and the clinicians will be asked to estimate survival time left with options being weeks, weeks to months, several months to years, indefinite number of years, or they may choose not to answer.

SECONDARY OUTCOMES:
Quality of life of patients and caregivers | Up to 6 months
  Quality of life is being assessed with a 10 question survey that inquires about overall well being, physical and emotional health, stressors, interaction, and mood. Depending on the question, a higher score may be worse (for example - how would you score your anxiety where 10 is worst; versus how would you score your emotional well being where 10 is worst). The minimum value for each question is 0 and the maximum is 10. This scale has been used in other studies with Beacon. A summary statistic for each patient will be developed depending on the individual responses. Full survey can be reviewed upon request.
Discordance in prognostic understanding over time | Up to 6 months.
  We will assess how patients, caregivers, and their clinicians differently understand prognosis of the patient in a longitudinal fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Alyx B Porter Umphrey, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Sharma A, Fruth B, Barrera C, Farfour HN, Mrugala MM, Edwin MK, Sloan JA, Porter AB. How much time do we have? Longitudinal perception of prognosis in newly-diagnosed high grade glioma patients and caregivers compared to clinicians. J Neurooncol. 2021 Apr;152(2):313-323. doi: 10.1007/s11060-021-03700-2. Epub 2021 Jan 23. PMID 33486637